CLINICAL TRIAL: NCT00351585
Title: A Double-blind, Placebo-controlled, Randomized, Parallel-group Study to Evaluate the Effects of Vildagliptin on the Maximum Insulin Secretion in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of Vildagliptin on the Maximum Insulin Secretion in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2344
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vildagliptin; Type 2 diabetes; Insulin secretion; Beta cell
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
Type 2 diabetes results when the body does not produce enough insulin to regulate blood sugar. This study is designed to measure the effect of vildagliptin on the maximum insulin secretion by the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for at least 6 months
* Patients whose diabetes is controlled by diet and exercise only or patients taking metformin
* BMI in the range 22-45
* Blood glucose criteria must be met

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes or diabetes resulting from pancreatic injury
* Cardiovascular complications as defined by the protocol
* Significant diabetic complications as defined by the protocol

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-07; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in maximal insulin secretory capacity at 12 weeks
Durability of this effect after a 2-week washout

SECONDARY OUTCOMES:
Change from baseline in beta-cell sensitivity to glucose at 12 weeks
Durability of this effect after a 2-week washout
Chance from baseline in glucagon secretion at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David D'Alessio, MD, Principal Investigator — University of Cincinnati

REFERENCES:
- [Derived] D'Alessio DA, Denney AM, Hermiller LM, Prigeon RL, Martin JM, Tharp WG, Saylan ML, He Y, Dunning BE, Foley JE, Pratley RE. Treatment with the dipeptidyl peptidase-4 inhibitor vildagliptin improves fasting islet-cell function in subjects with type 2 diabetes. J Clin Endocrinol Metab. 2009 Jan;94(1):81-8. doi: 10.1210/jc.2008-1135. Epub 2008 Oct 28. PMID 18957505